CLINICAL TRIAL: NCT03683264
Title: Forceps vs Vacuum. Rate of Levator Ani Muscle Avulsion: Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Valme (Other)
Responsible Party: Principal Investigator, José Antonio García Mejido, Principal Investigator, Hospital Universitario de Valme
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Forceps vs vacuum
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Birth Injuries; Pelvic Floor Disorders; Instrumental; Injury, Obstetric
MeSH Terms: conditions — Birth Injuries; Pelvic Floor Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum delivery (Other): Deliveries completed using vacuum instrumentation were performed by obstetricians with a minimum of five years' experience in obstetric practice. In terms of analgesia, epidural analgesia was used for intrapartum analgesia. The vacuum was a metal vacuum (Bird's cup 50 mm, 80 kPa) was used to perform fetal extraction. Traction was carried out during contraction, along with maternal push, at a rate of 2-3 tractions per contraction, and without associating Kristeller maneuver. The procedure was abandoned if, after three cup slides or 15 min, fetal extraction had not been successful. Selective episiotomy was carried out in vacuum delivery following Valme's University Hospital clinical practice guideline for instrumental deliveries.
  Interventions: Other: Ultrasound diagnosis of avulsion of the levator ani muscle
- Forceps delivery (Other): Deliveries completed using forceps instrumentation were performed by obstetricians with a minimum of five years' experience in obstetric practice. In terms of analgesia, epidural analgesia was used for intrapartum analgesia. The forceps used for the instrumentation was the forceps of Kielland. Traction was carried out during contraction, along with maternal push, at a rate of 2-3 tractions per contraction, and without associating Kristeller maneuver. The procedure was abandoned if, after three cup slides or 15 min, fetal extraction had not been successful. Selective episiotomy was carried out in VD following Valme's University Hospital clinical practice guideline for instrumental deliveries.
  Interventions: Other: Ultrasound diagnosis of avulsion of the levator ani muscle

INTERVENTIONS:
Other: Ultrasound diagnosis of avulsion of the levator ani muscle — In the multi-view ultrasound images, complete avulsion was defined as an abnormal insertion of LAM in the lower pubic branch identified in all three central slices, i.e. in the plane of minimal hiatal dimensions (PMD) and the 2.5 and 5.0mm slices cranial to this one. Levator hiatus measurements, transverse diameters, anteroposterior diameters and area were also determined in the same plane (PMD).

SUMMARY:
The main target is to determine levator ani muscle avulsion rate in vacuum delivery, comparing it to forceps delivery. As secondary goals, The aim to evaluate the difference in levator hiatus area among our study groups.

DETAILED DESCRIPTION:
Nulliparous women who were recruited for an initial evaluation from our maternity unit, Hospital Universitario Virgen de Valme. Participants were recruited prior to instrumentation at delivery and those meeting the inclusion criteria, being randomized into the two study groups (vacuum delivery or forceps delivery).

Deliveries completed using vacuum instrumentation were performed by obstetricians with a minimum of five years' experience in obstetric practice. In terms of analgesia, epidural analgesia was used for intrapartum analgesia. The forceps used for the instrumentation was the forceps of Kielland and the vacuum was a metal vacuum (Bird's cup 50 mm, 80 kPa) was used to perform fetal extraction. A suction cup was carefully placed over the flexion point, avoiding caput succedaneum, and rapid negative pressure was applied (over 2 min, until 0.6-0.8 kg/cm2 ). Traction was carried out during contraction, along with maternal push, at a rate of 2-3 tractions per contraction, and without associating Kristeller maneuver. The procedure was abandoned if, after three cup slides or 15 min, fetal extraction had not been successful. Selective episiotomy was carried out in VD following Valme's University Hospital clinical practice guideline for instrumental deliveries.

Obstetric parameters evaluated were: gestational age, labor induction, epidural analgesia, type of instrumentation, duration of second stage of labor, episiotomy and perineal tears. Fetal parameters studied after birth were: fetal sex, weight, head circumference, umbilical artery pH at birth, Apgar test result (at 1 and 5 min), presence of neonatal morbidity (cephalohaematoma, brachial plexus palsy, etc.), admission to neonatology department and neonatal mortality.

The sonographic evaluation was performed six months after delivery and was carried out by a single examiner, with more than five years experience exclusively in obstetric ultrasound, with specific training in 3/4D imaging and blinded to obstetric data relating to the delivery. A 500_ Toshiba Aplio (Toshiba Medical Systems Corp., Tokyo, Japan) ultrasound with an abdominal probe PVT-675MV 3D was used for the assessments. Images were acquired with patients in dorsal lithotomy position, placed on the gynecological examination table and under empty bladder conditions. The transducer was carefully placed on each patient's perineum, applying the minimal possible pressure. Three volume measurements were taken for each patient: at rest, with Valsalva maneuver and with maximum contraction. Then, offline analysis of ultrasound volumes was carried out. Analysis of ultrasound volumes was performed offline.

In the multi-view ultrasound images, complete avulsion was defined as an abnormal insertion of LAM in the lower pubic branch identified in all three central slices, i.e. in the plane of minimal hiatal dimensions (PMD) and the 2.5 and 5.0mm slices cranial to this one. Levator hiatus measurements, transverse diameters, anteroposterior diameters and area were also determined in the same plane (PMD).

ELIGIBILITY:
Inclusion Criteria:

* Delivery with forceps or vacuum
* Cephalic presentation
* Primiparity
* At term gestation (37-42 weeks)
* No prior pelvic floor corrective surgery
* Written informed consent

Exclusion Criteria:

* Pregnancies with severe maternal or fetal pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Compare the rate of levator ani muscle avulsion | at 6 months after randomisation
  To compare the rate of levator ani muscle avulsion in vacuum delivery versus the rate of the ate of levator ani muscle avulsion in forceps delivery.
  The avulsion is studied by 3D transperineal ultrasound, through the multiplanar study, including images at 2.5 mm from the plane of minimal dmensions. Avulsion was defined as the discontinuity of levator ani muscle fibres at their pubic insertion, which were identified in the three central slices of the multiplanar assessment.
Compare the levator ani muscle hiatus area (cm2) | at 6 months after randomisation
  To compare the levator ani muscle hiatus area (cm2) in vacuum delivery versus the levator ani muscle hiatus area (cm2) in forceps delivery.
  Levator hiatal dimensions can be determined on 3D ultrasound by identifying the plane of minimal dimensions, i.e., the plane which contains the minimal distance between the posterior symphyseal margin and the anterior margin of the levator ani loop immediately posterior to the anorectal angle.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio García Mejido, Principal Investigator — Hospital Universitario de Valme
Locations (1):
- Hospital Nuestra Señora de Valme, Seville, Spain